CLINICAL TRIAL: NCT03715556
Title: Prospective, Randomized and Blind Comparative Analysis Between Attraction of Restrict Control Versus Liberal Cardiac Frequency in Patients in Sepse With Atrial Fibrillation of High Ventricular Response
Brief Title: Control Versus Liberal Cardiac Frequency in Patients in Sepse With Atrial Fibrillation of High Ventricular Response
Acronym: FAARV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSInCor-FAARVSepsis
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Sepsis; Septic Shock; Atrial Fibrillation; Ventricular Fibrillation; Atrial Fibrillation Rapid
MeSH Terms: conditions — Sepsis; Shock, Septic; Atrial Fibrillation; Ventricular Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amiodarone (Active Comparator): Amiodarone (5 mg / kg EV in 30 minutes) will be the drug of choice in the Restricted group blinded to the principal investigator. If there is no reversal / control and there is no adverse event, a further dose of the same previously administered medicinal product will be performed within 30 minutes, amiodarone 3 mg / kg. After the second dose, continuous infusion of amiodarone at a dose of 900 mg in 24 hours will be initiated. Administration of the drug will be blinded within the first hour to the principal investigator.
  Interventions: Drug: Amiodarone; Drug: 0.9% physiological solution
- No intervention (Placebo Comparator): The Liberal group will receive only 0.9% physiological solution, also blinded to the principal investigator.
  Interventions: Drug: 0.9% physiological solution

INTERVENTIONS:
Drug: Amiodarone — Administration of the drug will be blinded within the first 48 hours for the principal investigator. Amiodarone (5 mg / kg EV in 30 minutes) will be the drug of choice in the Restricted group blinded to the principal investigator. If there is no reversal / control and there is no adverse event, a further dose of the same previously administered medicinal product will be performed within 30 minutes, amiodarone 3 mg / kg. After the second dose, continuous infusion of amiodarone at a dose of 900 mg in 24 hours will be initiated.
  Arms: Amiodarone
Drug: 0.9% physiological solution — Administration of 0.9% physiological solution.

SUMMARY:
Amiodarone is considered the medicine of choice in heart rate control in critically ill patients with atrial fibrillation with high ventricular response. However, a recent retrospective study showed a greater number of events in critical patients in whom there was an attempt to control versus in which there was no. Therefore, the prospective and randomized comparative use of amiodarone in this group of patients has not yet been described. The aim of this study was to evaluate the safety of the use of amiodarone (restricted group) versus placebo (liberal group) in heart rate control in atrial fibrillation with high ventricular response in patients with sepsis and vasopressor cardiovascular dysfunction. For this, a unicentric, randomized, blind and prospective study will be performed, in which the restrictive versus liberal strategy is performed in a comparative way. Hospital data (test results, medical evolutions complications) of patients will be analyzed to calculate safety and effectiveness. Expected results: The liberal strategy is superior to the restrictive strategy and causes fewer adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Permanent FA presence with FC> 110 bpm
* Presence of infection (any infectious outbreak)
* Cardiovascular dysfunction - need for vasopressor drugs (noradrenaline, adrenaline or vasopressin) to maintain SBP> 90 mmHg
* Signed consent form

Exclusion Criteria:

* Pregnancy
* Body mass index greater than 40 kg / m2
* Contraindication to the use of oral or parenteral anticoagulants
* Acute coronary syndrome
* Left ventricular ejection fraction <35%
* Valvular Heart Disease
* Contraindication to the use of amiodarone
* Child C cirrhosis
* Dialytic chronic renal insufficiency
* Chronic obstructive pulmonary disease
* Acute myocarditis
* Pulmonary thromboembolism
* Terminal neoplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Complications of safety outcomes | 48 hours
  Need for orotracheal intubation, Bradycardia requiring specific treatment or transvenous pacemaker, Confirmed embolic event, Need for association of another vasoactive drug or dose increase of already used vasoactive drug> 50% of initial, Cardiorespiratory arrest, Death

SECONDARY OUTCOMES:
Effectiveness in the control of the heart rate | 48 hours
  Comparison between the effectiveness in the control of the heart rate of AF among patients of the Restricted versus Liberal group. Effective control will be considered when the patient reaches heart rate <100 bpm

CONTACTS AND LOCATIONS:
Overall Officials: Mucio Tavares, MD, Principal Investigator — Unidade Clínica de Emergência
Locations (1):
- Instituto do Coração - HMFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided